CLINICAL TRIAL: NCT03261440
Title: Combined Cardiac, Pulmonary and Diaphragm Sonography for the Evaluation of Failure in Ventilation Weaning
Brief Title: Cardiac, Pulmonary and Diaphragm Sonography for the Early Diagnosis of the Different Etiologies Underlying Failure of Weaning From Mechanical Ventilation
Acronym: WEAN US
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: KLEIN 2016
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Mechanical Ventilation; Following Heart or Abdominal Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Weaning patients off ventilation in an ICU is sometimes difficult, because of three major inter-related etiologies: impaired lung, heart and diaphragm function. In this context, ultrasonography during tests to wean patients off ventilation could make it possible to diagnose cardiac dysfunction, a loss of pulmonary aeration or diaphragm dysfunction and thus reduce the number of failures at extubation.

The study will be carried out in 100 patients on mechanical ventilation following abdominal or heart surgery, who will have echocardiography, and pulmonary and diaphragm ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Patients on mechanical ventilation for at least 48 hours
* Age ≥ 60 years
* Patients who have undergone abdominal or heart surgery

Exclusion Criteria:

* Patients with a known neuromuscular disease
* Patients younger than 60 years
* Duration of mechanical ventilation <48h
* Non-surgical patients
* Patients with severe COPD

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on post-operative mechanical ventilation following heart or abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Echocardiography | At baseline
Lung ultrasonography | At baseline
Diaphragm ultrasonography | At baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Bouhemad B, Mojoli F, Nowobilski N, Hussain A, Rouquette I, Guinot PG, Mongodi S. Use of combined cardiac and lung ultrasound to predict weaning failure in elderly, high-risk cardiac patients: a pilot study. Intensive Care Med. 2020 Mar;46(3):475-484. doi: 10.1007/s00134-019-05902-9. Epub 2020 Jan 8. PMID 31915837